CLINICAL TRIAL: NCT03846752
Title: Complex Large-bore Radial PCI Trial Randomized Trial Reducing Access Site Complications With Slender Technology for Complex PCI
Brief Title: Complex Large-bore Radial Percutaneous Coronary Intervention (PCI) Trial
Acronym: Color
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maatschap Cardiologie Zwolle (Other)
Collaborators: Terumo Europe N.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9285; NL66831.075.18 (Registry Identifier: CCMO); 180716 (Other: Dutch ethical committe)
Record Dates: First submitted 2019-02-14; First posted 2019-02-20 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Complex Coronary Lesions
Keywords: Transradial Intervention; transfemoral intervention; PCI for complex coronary lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 7 Fr. radial access (Active Comparator): radial artery access for complex PCI
  Interventions: Procedure: radial artery access for complex PCI
- 7 Fr. femoral access (Active Comparator): femoral artery access for complex PCI
  Interventions: Procedure: femoral artery access for complex PCI

INTERVENTIONS:
Procedure: radial artery access for complex PCI — Complex PCI with access via radial artery using a 7 Fr. Glideslender sheath. PCI will be performed according to standard procedures and left to the discretion of the operator, however in case of stent placement the use of Ultimaster stents (Terumo) are highly recommended.
  Arms: 7 Fr. radial access
Procedure: femoral artery access for complex PCI — Complex PCI with access via femoral artery using a 7 Fr. standard femoral sheath . PCI will be performed according to standard procedures and left to the discretion of the operator, however in case of stent placement the use of Ultimaster stents (Terumo) are highly recommended.
  Arms: 7 Fr. femoral access

SUMMARY:
The COLOR trial is a Multicenter Randomized trial. Patients are eligible for study participation when PCI is indicated for complex coronary lesions. If patients comply with inclusion and exclusion and provide written informed consent they will be randomized in a 1:1 fashion between the two study treatments, (7 Fr. radial access with a Glideslender sheath or 7 Fr. femoral access with a standard femoral sheath) , in a 1:1 ratio.

DETAILED DESCRIPTION:
The COLOR trial is a Multicenter Randomized trial. Patients are eligible for study participation when PCI is indicated for complex coronary lesions. If patients comply with inclusion and exclusion and provide written informed consent they will be randomized in a 1:1 fashion between the two study treatments, (7 Fr. radial access with a Glideslender sheath or 7 Fr. femoral access with a standard femoral sheath) , in a 1:1 ratio.

During hospitalization (before discharge) the access site(s) will be checked for bleeding and vascular complications. All access sites should be checked for absent pulsations and hematomas and the size should be defined (length and width, cm) and accompanied complaints. Radial artery occlusion should be checked with the reverse Barbeau test. The femoral access site should be checked for murmurs and absence of pulsations. Ultrasound or Doppler of the access sites should be performed in those patients with suspected radial or femoral occlusion and the presence of other vascular complications, like (pseudo) aneurysms or arteriovenous (AV) fistula within 1 month.

Patient-reported extremity dysfunction will be evaluated at baseline (before the procedure) and 1-month follow-up. Upper extremity function will be evaluated with the Quick Disabilities of the Arm, Shoulder and Hand questionnaire (QuickDASH) and lower extremity function with Lower Extremity Functional Scale questionnaire (LEFS). The occurrence of Major Adverse Cardiac Events (MACE) will be evaluated at discharge and 1-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Use of 7 Fr guiding catheter is indicated for complex PCI, according to the expertise of the treating physician.
2. Age 18 years or older.

Exclusion Criteria:

1. Inability to obtain informed consent
2. contra-indication for radial or femoral access
3. Cardiogenic shock
4. ST-elevation myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is defined as BARC 2,3 and 5 (Bleeding Academic Research Consortium) bleeding or vascular complication related to the randomized access site (during hospitalization). | PCI procedure till patients is discharged from the hospital, with a maximum of 30 days
  The primary endpoint is defined as BARC 2,3 and 5 bleeding or vascular complication related to the randomized access site (during hospitalization).

SECONDARY OUTCOMES:
Non-access site related BARC 2,3 and 5 bleeding and/or vascular complications (hospitalization) | PCI procedure till patients is discharged from the hospital, with a maximum of 30 days
  Non-access site related BARC 2,3 and 5 bleeding and/or vascular complications (hospitalization)
MACE (hospitalization and 1-month) | PCI procedure till 30 days after PCI procedure
  MACE: Composite of death, myocardial infarction and repeat revascularization
Procedural success | during PCI procedure
  Successful PCI of the target lesion with a residual stenosis of less than 20%
procedural time | during PCI procedure
  Procedural time from puncture to end procedure (in minutes)
fluoroscopy time | during PCI procedure
  fluoroscopy time (in seconds)
contrast use | during PCI procedure
  Contrast volume used (in ml)
crossover rate | during PCI procedure
  Failure to complete the procedure through the randomized access site, requiring conversion from radial to femoral access or vice versa for procedure completion

CONTACTS AND LOCATIONS:
Overall Officials: Maarten A. Van Leeuwen, MD, Principal Investigator — Isala
Locations (12):
- Belgium (3):
  - ZNA Middelheim, Antwerp
  - CHU Charleroi, Charleroi
  - Ziekenhuis Oost Limburg, Genk
- Elisabeth Krankenhaus, Essen, Germany
- Netherlands (6):
  - Isala, Zwolle, Overijssel
  - Noordwest Ziekenhuisgroep, Alkmaar
  - OLVG, Amsterdam
  - VUMC, Amsterdam
  - Catharina Ziekenhuis Eindhoven, Eindhoven
  - RadboudUMC, Nijmegen
- University Hospital Geneva, Geneva, Switzerland
- Frimley Health NHS Foundation Trust, Surrey, Camberley, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The availability of individual participant data will be separately decided for each request by the PI of the study. The sponsor will have to agree before publication.
  All data that is required to minimally fulfill the request will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Data is available after publication of final specific subgroup analyses, no predetermined end-date
Access Criteria: Proposals should be directed to the PI of the study (m.a.h.van.leeuwen@isala.nl). To gain access, data requestors will need to sign a data transfer agreement.

REFERENCES:
- [Derived] Meijers TA, Nap A, Aminian A, Dens J, Teeuwen K, van Kuijk JP, van Wely M, Schmitz T, Bataille Y, Kraaijeveld AO, Roolvink V, Hermanides RS, Braber TL, van Royen N, van Leeuwen MAH. ULTrasound-guided TRAnsfemoral puncture in COmplex Large bORe PCI: study protocol of the UltraCOLOR trial. BMJ Open. 2022 Dec 1;12(12):e065693. doi: 10.1136/bmjopen-2022-065693. PMID 36456007
- [Derived] Meijers TA, Aminian A, van Wely M, Teeuwen K, Schmitz T, Dirksen MT, Rathore S, van der Schaaf RJ, Knaapen P, Dens J, Iglesias JF, Agostoni P, Roolvink V, Lemmert ME, Hermanides RS, van Royen N, van Leeuwen MAH. Extremity Dysfunction After Large-Bore Radial and Femoral Arterial Access. J Am Heart Assoc. 2022 Jan 18;11(2):e023691. doi: 10.1161/JAHA.121.023691. Epub 2022 Jan 13. PMID 35023343
- [Derived] Meijers TA, Aminian A, van Wely M, Teeuwen K, Schmitz T, Dirksen MT, Rathore S, van der Schaaf RJ, Knaapen P, Dens J, Iglesias JF, Agostoni P, Roolvink V, Hermanides RS, van Royen N, van Leeuwen MAH. Randomized Comparison Between Radial and Femoral Large-Bore Access for Complex Percutaneous Coronary Intervention. JACC Cardiovasc Interv. 2021 Jun 28;14(12):1293-1303. doi: 10.1016/j.jcin.2021.03.041. Epub 2021 May 18. PMID 34020929
- [Derived] Meijers TA, Aminian A, Teeuwen K, van Wely M, Schmitz T, Dirksen MT, van der Schaaf RJ, Iglesias JF, Agostoni P, Dens J, Knaapen P, Rathore S, Ottervanger JP, Dambrink JE, Roolvink V, Gosselink ATM, Hermanides RS, van Royen N, van Leeuwen MAH. Complex Large-Bore Radial percutaneous coronary intervention: rationale of the COLOR trial study protocol. BMJ Open. 2020 Jul 20;10(7):e038042. doi: 10.1136/bmjopen-2020-038042. PMID 32690749